CLINICAL TRIAL: NCT06005961
Title: A Randomised Controlled Trial of Module-Based Psychological (MBP) Intervention for Young People with Mental Distress in Hong Kong
Brief Title: Module-Based Psychological (MBP) for Community Youths
Acronym: MBP_RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Christy Lai-ming Hui, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBP_intervention
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorder; Depressive Symptoms; Anxiety Symptoms
Keywords: randomised controlled trial; module-based psychological intervention; youths; mental distress
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBP intervention arm (Active Comparator): The MBP intervention has two modules: the core and the tailor-made modules. The core module focuses on emotional management, while the five tailor-made modules include anxiety management, mood and depression management, anger management, sleeping well, and managing self-expectation and compassion.
  Interventions: Behavioral: Module-Based Psychological (MBP) Intervention
- Waitlist control arm (Other): Participants allocated to the waitlist control group will wait for 6 plus 4 weeks before receiving the MBP intervention.
  Interventions: Behavioral: Module-Based Psychological (MBP) Intervention

INTERVENTIONS:
Behavioral: Module-Based Psychological (MBP) Intervention — Participants will receive one core module related to emotional management and maximum two tailor-made modules according to the participant's needs. Each weekly session lasts for 1 hours. The core module will last for 6 weeks and the tailor-made modules will last for 3 - 4 weeks.

SUMMARY:
This waitlist, randomised controlled trial (RCT) aims to examine the effectiveness of the Module-Based Psychological (MBP) intervention in reducing mental distress for youths aged 12-30 years in Hong Kong. The participants randomised to the MBP group will receive 4-7 sessions of MBP (in 6 to 10 weeks) in an individual format delivered by frontline social or youth workers trained by professional clinicians. The waitlist control group will receive the same intervention after 6 weeks of waiting plus a 1-month follow-up period. The MBP is designed to improve the youths' abilities/skills in handling moods for better emotional management. Written informed consent will be signed by participants or their parents/guardians if they are under the age of 18.

DETAILED DESCRIPTION:
This randomised controlled trial (RCT) aims to examine the effectiveness of the Module-Based Psychological (MBP) intervention in reducing mental distress for youths in Hong Kong. This intervention study will be delivered in an individual format for 4 sessions of core module in 6 weeks plus/minus 2-3 sessions of tailored-made module in 3-4 weeks by frontline social or youth workers trained by professional clinicians. It is designed to improve the youths' abilities and skills in handling moods for better emotional management. The MBP intervention has two modules: core and tailor-made modules. The core module focuses on emotional management, while the five tailor-made modules include anxiety management, mood and depression management, anger management, sleeping well, and managing self-expectation and compassion. The tailor-made modules will be assigned to youths according to their needs. While the clinical outcome of the MBP is evaluated, its cost-effectiveness is also of particular concern. Planned interim analyses are built into the project for the sake of evaluation of the collected data from the ongoing trial, in which the primary research question is addressed and which has the potential to modify the conduct of the study. It is hypothesised that the youths who have received MBP intervention will demonstrate a greater reduction in mental distress, depressive symptoms, and anxiety symptoms compared to the youths in the waitlist control group. Besides, the MBP intervention will be more cost-effective than waiting.

ELIGIBILITY:
Inclusion Criteria:

1. LevelMind@JC users aged from 12-30
2. Reported at-least mild mental distress
3. Have sufficient proficiency in Chinese to understand verbal instructions
4. Able to give informed consent

Exclusion Criteria:

1. Known diagnosis of intellectual disability
2. Known diagnosis of organic brain disorder
3. Known psychiatric diagnosis within two years
4. Current substance abuse
5. Receiving any psychiatric treatments or structural psychological therapies such as cognitive behavioural therapy, mentalisation-based therapy and low-intensity online intervention, narrative therapy, mindfulness, and art-informed therapy
6. Current or active suicidal ideation or attempts

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
General mental distress | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the Kessler Psychological Distress Scale, 6-item version (K6). The total K6 score ranges from 0 to 24, with higher scores indicating a greater distress level.
Depressive symptoms | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the 7-item Depression Subscale of the Depression, Anxiety, and Stress Scale, 21-item version (DASS-D).
  The total score ranges from 0-42, with higher scores indicating greater severity of depressive symptoms.
Anxiety symptoms | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the 7-item Anxiety Subscale of the Depression Anxiety and Stress Scale 21-item version (DASS-A) The total score ranges from 0-42, with higher scores indicating greater severity of anxiety symptoms.
Functioning | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the Social and Occupational Functioning Assessment Scale (SOFAS).
  The score ranges from 0-100, with higher scores indicating better social and occupational functioning related to physical and mental health.

SECONDARY OUTCOMES:
Health-related quality of life | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the 12-Item Short Form Health Survey (SF-12). The derived index score ranges from 0-100, with higher scores indicating better physical and mental health functioning.
Self-compassion | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the 12-item Self-Compassion Scale (SCS). The total score ranges from 5-60, with higher scores indicating better self-compassion.
Self-efficacy | baseline (T0), post-treatment (6-week, T1), and follow-up (9 week, T2)
  Measured using the 10-item General Self-Efficacy Scale (GSE). The total score ranges from 10 and 40, with higher scores indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Christy Lai-ming Hui, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No